CLINICAL TRIAL: NCT01951261
Title: Early Assisted Discharge With Generic Community Nursing and Pulmonary Physicians vs Telemonitoring at Home for Chronic Obstructive Pulmonary Disease Exacerbations
Brief Title: Early Assisted Discharge for COPD Exacerbations With Telemonitoring.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. López Viña (Other)
Responsible Party: Sponsor-Investigator, Dr. López Viña, Investigator, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TELEMEDCOPD
Record Dates: First submitted 2013-09-03; First posted 2013-09-26 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: COPD Exacerbation
Keywords: Telemonitoring; COPD; Home care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telemonitoring and telephone control (Active Comparator): Early discharge from hospital with telemonitoring, telephone control and three nurse scheduled visits.
  Interventions: Procedure: Telemonitoring and telephone control
- home care (No Intervention): Early discharge from hospital with home care provided by hospital respiratory nurses and pulmonologists (daily visits).

INTERVENTIONS:
Procedure: Telemonitoring and telephone control — Early assisted discharge from hospital due to an exacerbation of chronic obstructive pulmonary disease, with telemonitoring of vitals signs (oxygen saturation, heart rate, respiratory rate, blood pressure, temperature and electrocardiogram)and telephone control dairy (morning, evening)by the pulmonologist.
  Arms: telemonitoring and telephone control

SUMMARY:
To determine if an early assisted discharge program for acute exacerbations of COPD (AECOPD), with telemonitoring and telephone control, is equally effective and more efficient in terms of use of health care resources, that a home care provided by hospital respiratory nurses and pulmonologists.

DETAILED DESCRIPTION:
This study seeks to improve the health of patients with AECOPD by home care after discharge from the Hospital using the technology of the information and the communication. The investigators want evaluate the efficiency, satisfaction (patients, keepers) and effectiveness of a program of early discharge with home care in patients with AECOPD with telemonitoring and telephone control, in relation to the traditional protocol of home care based on nurse and pulmonologist visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hospital with COPD exacerbation
* No concomitant serious unstable diseases
* Without fever in 48 hours
* Aerosol treatment at the most every 6 hours
* Treatment with glucocorticoid intravenous < 40 mg twice a day
* A thoracic radiograph without new disease
* Subjective improvement of the patient
* Familiar suitable environment

Exclusion Criteria:

* Neoplasias and other chronic diseases in terminal situation
* Alcoholism
* Intravenous medication
* Disability to understand and take part in the program
* Admitted to intensive care unit (ICU) or non invasive mechanical ventilation during the exacerbation
* Unstability hemodynamic
* To be an institutionalized patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antolín Lopez Viña, physician, Study Director — Hospital Puerta de Hierro; Antolín Lopez Viña, MD, Principal Investigator — Hospital Puerta de Hierro
Locations (1):
- Universitary Hospital Puerta de Hierro., Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Share All of the individual participant data collected during the trial, after identification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Proposals should be directed to drapat1@yahoo.es. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Care: Early discharge from hospital with home care provided by hospital respiratory nurses and pulmonologists (dairy visits).
Period: Overall Study
Arm/Group | Telemonitoring and Telephone Control | Home Care
Started | 58 | 58
Discontinued | 9 (2-readmission when was at home 1-monitor failure 1-new home hospitalitation 4-missing 1-death) | 6 (2-readmission when was at home 1-new home hospitalitation 3-missing)
Completed | 49 | 52
Not Completed | 9 | 6
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telemonitoring and Telephone Control | Home Care | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8) | 70 (8) | 69 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 23 | 36
  Male | 45 | 35 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index (BMI) (Mean (Standard Deviation) [Mean (Standard Deviation); unit: Kg/m^2] | 27.1 (4) | 26.5 (4) | 26.8 (4)

OUTCOME MEASURES:

1. Primary Outcome: Time Until the First Exacerbation
Description: Time until the first exacerbation is the time that patient is stable before a new exacerbation and meaning a good control of the disease.
Time Frame: Change from stable to exacerbation the first time at 6 month
Population: The overall number of participants analyzed is not consistent with numbers provided in any of the rows in the participant flow module, because in the telemedicine group and the home care group, patients who readmission were not included, nor was the patient in whom the monitor did not work.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Telemonitoring and Telephone Control | Home Care
Number analyzed (Participants) | 54 | 55
days | 47 [19 to 102] | 48 [23 to 120]
Statistical Analysis 1: Comparison: Telemonitoring and Telephone Control vs Home Care; Test type: Non-Inferiority — sample size calculation was made, considering it appropriate to set a limit of non-inferiority with respect to the main variable of 1.2 months (36 days), the study being lower if it will have exacerbation before this period of time, with a follow-up of 6 months, It was required to include a sample of 58 patients per group for a potency of 80% and a significance level of 5%; p < 0.05, Log Rank — The reported p-value was calculated.Statistical analysis of the main variable was performed using the Kaplan-Meier method and log-rank test

2. Secondary Outcome: SATISFAD 10
Description: Instrument that evaluates satisfaction with home care services in a self-administered. The score ranges from 0 to 30, with the worst value being zero and the best value being 30.
Time Frame: Participants will be followed for the duration home care, an expected average of 7 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Telemonitoring and Telephone Control | Home Care
Number analyzed (Participants) | 37 | 42
score on a scale | 30 [29 to 30] | 30 [27 to 30]

3. Secondary Outcome: State-Trait Anxiety Inventory (STAI)
Description: The structure of the scale resulting from the combination of item polarity dimensions and the original two factors (State and Trait Anxiety).
  Minimum value 0, maximum value 120. Lower score indicates higher anxiety.
Time Frame: Participants will be followed for the duration of home care, an expected average of 7 days
Population: Not all study participants completed the test, so it does not correspond to the number of the flow chart.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Telemonitoring and Telephone Control | Home Care
Number analyzed (Participants) | 44 | 44
score on a scale
  State | 15 [10 to 26] | 17 [12 to 25]
  Trait | 20 [15 to 26] | 23 [17 to 27.5]

4. Secondary Outcome: Percentage of Participants With Medication Adherence Assessed Using Morinsky-Green-Levine Test
Description: Consists of a series of 4 contrasting questions with answers dichotomous yes / no, reflecting the patient's behavior regarding compliance with medication. They are intended to assess whether the patient adopts correct attitudes regarding treatment for his illness; it is assumed that if attitudes they are incorrect the patient is non-compliant.
Time Frame: Participants will be followed for the duration of home care up 24 weeks
Population: Not all study participants completed the test, so it does not correspond to the number of the flow chart.
Measure: Number; unit: percentage of adherents
Arm/Group | Telemonitoring and Telephone Control | Home Care
Number analyzed (Participants) | 44 | 41
percentage of adherents
  Initial | 77 | 78
  At 6 month | 86 | 87

5. Secondary Outcome: Monitoring Compliance
Description: It represents the compliance of the patients with respect to the sending of constants through the telemedicine monitor that should be (following the protocol) at least twice a day. The patient was considered compliant if he sent the constant at least 2 twice a day or non-compliant otherwise.
Time Frame: Participants will be followed for the duration of home care, an expected average of 7 days
Population: In the home care group, patients did not send constants. Data from 55 patients were analyzed (2 readmissions and one patient in which the monitor failed were not included in the analysis)
Measure: Mean (Standard Deviation); unit: sending of constant
Arm/Group | Telemonitoring and Telephone Control | Home Care
Number analyzed (Participants) | 55 | 0
sending of constant | 2.23 (1) |

6. Secondary Outcome: Number of Home Visits
Time Frame: Participants will be followed for the duration of home care, an expected average of 7 days
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Telemonitoring and Telephone Control | Home Care
Number analyzed (Participants) | 56 | 57
visits | 3.8 (1) | 5.1 (2)

7. Secondary Outcome: COPD Assessment Test (CAT)
Description: It's a simple questionnaire for assessing and monitoring COPD. It quantifies chronic obstructive pulmonary disease (COPD) impact in routine practice to aid health status assessment.
  It's self-administered in 2 min. It consists of 8 items that measure aspects of cough, expectoration, chest tightness, dyspnea, domestic activities, self-confidence, sleep and energy. Each section is scored from 0 to 5 and therefore a maximum of 40 points can be obtained; a higher score indicates a greater negative impact of COPD. Significant clinical changes correspond to a variation of 2 points or more.
Time Frame: Participants will be followed for the duration of home care and up to 4 weeks
Population: Not all study participants completed the test, so it does not correspond to the number of the flow chart.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Telemonitoring and Telephone Control | Home Care
Number analyzed (Participants) | 49 | 49
score on a scale
  Initial | 10 [7 to 15] | 15 [9 to 21]
  At first month | 8 [5 to 15] | 8 [4.5 to 11]

ADVERSE EVENTS:
Time Frame: During home follow-up until 6 months after the discharge.
Description: All adverse events caused the patient to be hospitalized.
Arm/Group | Telemonitoring and Telephone Control | Home Care
All-Cause Mortality (participants affected / at risk) | 1/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 2/58 | 2/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telemonitoring and Telephone Control (N=58) | Home Care (N=58)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
rapid atrial fibrillation (Cardiac disorders) | 1 | 0
necrotizing pneumonia. (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pain secondary to vertebral crushing (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-02-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT01951261/Prot_SAP_000.pdf
  • Informed Consent Form (2012-02-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT01951261/ICF_001.pdf